CLINICAL TRIAL: NCT05484661
Title: Mechanisms to Reduce Mental and Physical Fatigue Following Exercise Training in Older Adults
Acronym: BCAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Monica Serra, Associate Professor, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20220493H
Record Dates: First submitted 2022-07-28; First posted 2022-08-02 (Actual); Results first posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-10

CONDITIONS: Fatigue; Aging
Keywords: Branched Chain Amino Acids; Exercise
MeSH Terms: conditions — Fatigue; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise + BCAA (Experimental): Exercise will include a 3x/wk for eight weeks exercise protocol is designed to provide a high-volume, moderate-intensity whole body training stimulus. BCAA will include ~7-10 g of BCAAs (100 mg/kg) daily for eight weeks.
  Interventions: Dietary Supplement: BCAA
- Exercise + Placebo (Placebo Comparator): Exercise will include a 3x/wk for eight weeks exercise protocol is designed to provide a high-volume, moderate-intensity whole body training stimulus. Placebo will include ~7-10 g of maltodextrin (100 mg/kg) daily for eight weeks.
  Interventions: Dietary Supplement: BCAA

INTERVENTIONS:
Dietary Supplement: BCAA — Participants will participate in high-volume, moderate-intensity exercise 3x/week and consume either a placebo or BCAA (~7-10 g of BCAAs (100 mg/kg) daily for eight weeks.

SUMMARY:
Fatigue is a strong predictor of negative health outcomes in older adults. The research in this study will compared the effects of 8-weeks of branched chain amino acids (BCAAs: dietary supplements commonly taken to improve muscle growth and exercise performance) added to exercise on fatigue compared to exercise with a placebo (an inactive, harmless substance). BCAAs could have an impact on improving fatigue common in older adults, especially when exercising.

DETAILED DESCRIPTION:
Thirty participants will be asked to participate in this research study. They will be randomized (like a flip of a coin) to exercise + a placebo or exercise + BCAAs for 8 weeks. We would like to examine the effects of the 8-week exercise + dietary supplement program on body composition (fat and muscle), physical activity habits, fatigue, and physical performance (such as walking and strength). We would also like to assess whether these outcomes are controlled by changes in markers (kynurenine metabolites) in the skeletal muscle and blood.

ELIGIBILITY:
Inclusion Criteria:

* Fatigue (participants reporting ≥3 on a 1-10 scale)
* Lack of menses for at least one year for women
* BMI 20-50 kg/m2
* Untrained with regard to structured exercise training (is not currently training more than 2x/week)

Exclusion Criteria:

* Taking an anticoagulant medication that is unable to be discontinued before biopsies
* Allergic to lidocaine
* Neurologic, musculoskeletal, or other condition that limits subject's ability to complete study physical assessments or training
* Hepatic (LFTs >2.5xWNL), renal (eGFR<45), , and uncontrolled psychiatric disease
* Cognitive impairment
* Uncontrolled depression
* Any disease or condition considered to be exclusionary based on the clinical opinion and discretion of the principal investigator

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Robbins RN, Cortes T, O'Connor JC, Jiwani R, Serra MC. The Influence of Branched-Chain Amino Acid Supplementation on Fatigue and Tryptophan Metabolism After Acute and Chronic Exercise in Older Adults: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2023 Nov 1;12:e52199. doi: 10.2196/52199. PMID 37910166

RESULTS

PARTICIPANT FLOW:
Groups:
- Exercise + BCAA: Exercise will include a 3x/wk for eight weeks. Exercise protocol is designed to provide a high-volume, moderate-intensity whole body training stimulus. BCAA will include ~7-10 g of BCAAs (100 mg/kg) daily for eight weeks.
Period: Overall Study
Arm/Group | Exercise + BCAA | Exercise + Placebo
Started | 10 | 10
Completed | 9 | 10
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise + BCAA | Exercise + Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.4 (3.6) | 70.0 (3.1) | 70.0 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 9 | 12
  Male | 7 | 1 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 10 | 9 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Fatigue
Description: Participants will complete the Fatigue Assessment Scale questionnaire (Total scores can range from 10, indicating the lowest level of fatigue, to 50, denoting the highest)
Time Frame: change from baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: change in fatigue severity score
Arm/Group | Exercise + BCAA | Exercise + Placebo
Number analyzed (Participants) | 9 | 10
change in fatigue severity score | -5.6 (4.0) | -4.1 (3.1)

ADVERSE EVENTS:
Time Frame: Up to 8 weeks
Arm/Group | Exercise + BCAA | Exercise + Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-11): https://cdn.clinicaltrials.gov/large-docs/61/NCT05484661/Prot_SAP_000.pdf